CLINICAL TRIAL: NCT06819683
Title: The Validation of Minimally Invasive Oxygen Nanosensor Technology to Quantify Mitochondrial Function in Human Muscle
Brief Title: Validation of Nanosensor Oxygen Measurement
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-019820; W81XWH2210590 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2025-02-04; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: MItochondrial Myopathies; Mitochondrial Disease
MeSH Terms: conditions — Mitochondrial Myopathies; Mitochondrial Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Affected Mitochondrial Myopathy (MM) Cases (Experimental): Key eligibility criteria for Mitochondrial Myopathy (MM) cases includes physically-capable adults (male and females, ages 18 to 65 years, inclusive) with genetically-confirmed MM with predominant symptoms of myopathy as expressed by exercise intolerance and muscle weakness and fatigue.
  Interventions: Device: Nanosensor
- Healthy Controls (Active Comparator): Adult healthy volunteers will be individually matched with corresponding Mitochondrial Myopathy cases based on age, biological sex, and body mass index.
  Interventions: Device: Nanosensor

INTERVENTIONS:
Device: Nanosensor — The purpose of the study is to test a device called a "nanosensor", which measures oxygen levels (a proxy of mitochondrial function) in muscle. The nanosensor has not been tested in humans nor has it been approved by the FDA. The study nanosensor measures 1.8 mm width x 6 mm length x 0.3 mm depth. Placement of the sterilized nanosensor involves a small incision for manual placement of the nanosensor in muscle forearm tissue.

SUMMARY:
Past mitochondrial disease treatment studies have been unsuccessful in determining treatment efficacy, and a major factor has been the lack of validated biomarkers in mitochondrial myopathy (MM). There is currently a growing number of potential new treatments to be tested through MM clinical intervention trials, which has created a pressing need for quantitative biomarkers that reliably reflect MM disease severity, progression, and therapeutic response. The purpose of the study is to measure the efficacy of an electrochemical oxygen nanosensor to measure in vivo mitochondrial function in human muscle tissue, and its ability to discriminate MM patients from healthy volunteers. The data and results from this nanosensor study may contribute to current and future research, including improved diagnostic and therapeutic approaches for patients with mitochondrial disease.

DETAILED DESCRIPTION:
This is an investigational device clinical trial. Mitochondrial Myopathy (MM) cases and healthy volunteers will undergo nanosensor muscle oxygen measurement in exercised (dominant) forearm muscle during handgrip exercise.

After placement of the nanosensor in the forearm under local anesthesia, the primary outcome measure is nanosensor-muscle oxygen levels. The secondary outcome measure is an assessment of pain.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria for Healthy Controls

  1. Males and females, between the ages of 18 and 65 years, inclusive
  2. Provide informed consent for study participation; able to understand and complete the protocol
  3. Able to ambulate independently
  4. Able to perform bicycle ergometry

Inclusion Criteria for Mitochondrial Myopathy (MM) Cases

1. Males and females, between the ages of 18 and 65 years, inclusive
2. Provide informed consent for study participation; able to understand and complete the protocol
3. Genetically-confirmed MM as defined by a diagnosis of primary mitochondrial disease (PMD) with predominant symptoms of myopathy as expressed by exercise intolerance and muscle weakness and fatigue.
4. Previously enrolled (or will enroll) in Children's Hospital of Philadelphia (CHOP) Institutional Review Board (IRB) study #08-006177 (Falk, PI) or CHOP IRB #16-013364 (Zolkipli, PI)
5. Able to ambulate independently
6. Able to perform bicycle ergometry

Exclusion Criteria:

Subjects will be excluded if any of the following apply:

1. Unable to provide informed consent and complete all study procedures, including ergometry
2. Non-ambulatory or unable to ambulate independently
3. Pregnant
4. Within 1 month of a recent hospital admission due to acute illness
5. Have severe cardiac disease as defined by an ejection fraction of less than 35% and New York Heart Association Functional Classification Class III; or severe pulmonary disease as defined by the need for supplemental O2 therapy or daytime ventilatory support
6. Have a tracheostomy
7. Have a known bleeding disorder and/or family history (first-degree relative) with a known bleeding disorder
8. Daily intake of aspirin or any other anti-platelet therapy which cannot be temporarily discontinued for medical reasons
9. a) Have known or suspected congenital or acquired immune deficiency; b) concurrent use of immunosuppressive drugs, including corticosteroids; c) past history of recurrent (more than 6 times per year) severe (required hospitalization) skin or soft tissue infections; d) history of infection or delayed wound healing after surgery or biopsy; e) known history of neutropenia with absolute neutrophil count less than 500/mm3
10. Undergo chronic steroid treatment as defined by daily oral intake (for more than 1 month) or have existing untreated endocrinopathies, such as hypothyroidism that caused acquired myopathy
11. Prone to hypertrophic scars and keloids
12. Have any other known inherited myopathy, such as Duchenne muscular dystrophy or congenital myopathy
13. Known allergy to lidocaine
14. Have a cognitive impairment that may prevent the ability to complete study procedures
15. Unable to comply with the requirements of the study protocol and/or unsuitable for the study for any reason, in the opinion of the principal investigator
16. Individuals from vulnerable populations (e.g., prisoners/detainees)
17. Participants who are unable to speak and/or read English (as participants will be required to be proficient to complete study procedures)
18. Employed by the U.S. Department of Defense, including U.S. military personnel

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Nanosensor-muscle oxygen (Torr) levels during handgrip exercises | before, during and after handgrip exercise up to 4 hours or up to 40 days after the screening visit
  Nanosensor-muscle oxygen (Torr) levels will be measure in the (dominant) forearm muscle during handgrip exercises and correlated to the standard measure of venous oxygenation (VO2) levels using standard clinical indirect calorimetry as a measure of tissue oxygen consumption. This data will be reported as the Torr value at each time point during measurement.
Nanosensor-muscle oxygen (Torr) levels post Cardiopulmonary Exercise Testing (CPET) | After CPET exercise up to 1-hour
  Nanosensor-muscle oxygen (Torr) levels after cardiopulmonary exercise testing (CPET) will be measured in the (dominant) forearm muscle by comparing exercised muscle oxygen levels to the venous oxygen (VO2max) levels recorded during the CPET exercise. This data will be reported as the Torr value at each time point during measurement.

SECONDARY OUTCOMES:
Self-reported pain level assessment | up to 40 days after the screening visit
  After the exercise procedure, participants will self-report the level of pain/discomfort with the validated Wong-Baker Faces Pain Rating Scale and Numerical Rating Scale. The Wong-Baker Faces Pain Rating Scale is a tool used to assess pain levels in young children by presenting using a combination of faces, numbers, and words to help the participant effectively communicate the severity of their physical pain. The scale includes a happy face indicating 0="no hurt" to a crying face signifying 10="hurts worst." The NRS is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable." All subjects will respond to both surveys.
Patient Satisfaction | After study procedures are completed (approximately day 40)
  Patient satisfaction will be measured by participants completing the Post-operative Patient Satisfaction Survey. The survey consists of one question to gauge self-reported insight on their overall experience. Responses note the experience was "Agreeable", "Neither pleasant nor unpleasant", "Slightly uncomfortable", "Disagreeable", or "Traumatic".
Self-reported fatigue | After study procedures are completed (approximately day 40)
  After the exercise period, participants will self-report the level of fatigue as a measure of disease burden using the Modified Fatigue Impact Scale (MFIS). This scale includes 9 questions regarding subject's fatigue symptoms and how it impacts their life. Answers range from "Strongly Agree" to "Strongly Disagree" with 7 answer choices for each question.

CONTACTS AND LOCATIONS:
Overall Officials: Zarazuela Zolkipli-Cunningham, MBChB, MRCP, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No